CLINICAL TRIAL: NCT01839916
Title: Pilot Study of Prophylactic Dose-Escalation Donor Lymphocyte Infusion After T Cell Depleted Allogeneic Stem Cell Transplant in High Risk Patients With Hematologic Malignancies
Brief Title: Donor T Cells After Donor Stem Cell Transplant in Treating Patients With Hematologic Malignancies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-1191; NCI-2013-00782 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2013-04-22; First posted 2013-04-25 (Estimated); Results first posted 2019-08-07 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2019-06

CONDITIONS: Accelerated Phase Chronic Myelogenous Leukemia; Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Del(5q); Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(15;17)(q22;q12); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Adult Nasal Type Extranodal NK/T-cell Lymphoma; Anaplastic Large Cell Lymphoma; Angioimmunoblastic T-cell Lymphoma; Blastic Phase Chronic Myelogenous Leukemia; Childhood Burkitt Lymphoma; Childhood Chronic Myelogenous Leukemia; Childhood Diffuse Large Cell Lymphoma; Childhood Immunoblastic Large Cell Lymphoma; Childhood Myelodysplastic Syndromes; Childhood Nasal Type Extranodal NK/T-cell Lymphoma; Chronic Phase Chronic Myelogenous Leukemia; Cutaneous B-cell Non-Hodgkin Lymphoma; de Novo Myelodysplastic Syndromes; Extranodal Marginal Zone B-cell Lymphoma of Mucosa-associated Lymphoid Tissue; Hepatosplenic T-cell Lymphoma; Intraocular Lymphoma; Nodal Marginal Zone B-cell Lymphoma; Noncutaneous Extranodal Lymphoma; Peripheral T-cell Lymphoma; Post-transplant Lymphoproliferative Disorder; Previously Treated Myelodysplastic Syndromes; Recurrent Adult Acute Lymphoblastic Leukemia; Recurrent Adult Acute Myeloid Leukemia; Recurrent Adult Burkitt Lymphoma; Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Adult Diffuse Mixed Cell Lymphoma; Recurrent Adult Diffuse Small Cleaved Cell Lymphoma; Recurrent Adult Grade III Lymphomatoid Granulomatosis; Recurrent Adult Hodgkin Lymphoma; Recurrent Adult Immunoblastic Large Cell Lymphoma; Recurrent Adult Lymphoblastic Lymphoma; Recurrent Adult T-cell Leukemia/Lymphoma; Recurrent Childhood Acute Lymphoblastic Leukemia; Recurrent Childhood Acute Myeloid Leukemia; Recurrent Childhood Anaplastic Large Cell Lymphoma; Recurrent Childhood Grade III Lymphomatoid Granulomatosis; Recurrent Childhood Large Cell Lymphoma; Recurrent Childhood Lymphoblastic Lymphoma; Recurrent Childhood Small Noncleaved Cell Lymphoma; Recurrent Cutaneous T-cell Non-Hodgkin Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Marginal Zone Lymphoma; Recurrent Mycosis Fungoides/Sezary Syndrome; Recurrent Small Lymphocytic Lymphoma; Recurrent/Refractory Childhood Hodgkin Lymphoma; Refractory Chronic Lymphocytic Leukemia; Refractory Hairy Cell Leukemia; Relapsing Chronic Myelogenous Leukemia; Secondary Myelodysplastic Syndromes; Small Intestine Lymphoma; Splenic Marginal Zone Lymphoma; T-cell Large Granular Lymphocyte Leukemia; Testicular Lymphoma; Waldenström Macroglobulinemia
MeSH Terms: conditions — Leukemia, Myeloid, Accelerated Phase; Congenital Abnormalities; Lymphoma, Extranodal NK-T-Cell; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Blast Crisis; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Leukemia, Myeloid, Chronic-Phase; Intraocular Lymphoma; Lymphoma, B-Cell, Marginal Zone; Lymphoma, T-Cell, Peripheral; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Lymphoma, Non-Hodgkin; Hodgkin Disease; Lymphoma, Large-Cell, Immunoblastic; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Dendritic Cell Sarcoma, Interdigitating; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Mycosis Fungoides; Sezary Syndrome; Leukemia, Lymphocytic, Chronic, B-Cell; Recurrence; Leukemia, Hairy Cell; Leukemia, Large Granular Lymphocytic; Waldenstrom Macroglobulinemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (DLI) (Experimental): Patients receive DLI IV. Treatment repeats every 4-8 weeks for 5 doses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: therapeutic allogeneic lymphocytes; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: therapeutic allogeneic lymphocytes — Given IV
  Other Names: ALLOLYMPH
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This pilot phase II trial studies how well giving donor T cells after donor stem cell transplant works in treating patients with hematologic malignancies. In a donor stem cell transplant, the donated stem cells may replace the patient's immune cells and help destroy any remaining cancer cells (graft-versus-tumor effect). Giving an infusion of the donor's T cells (donor lymphocyte infusion) after the transplant may help increase this effect.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the feasibility of escalating dose regimen (EDR) donor lymphocyte infusion (DLI) as measured by the proportion of patients who receive at least one DLI.

SECONDARY OBJECTIVES:

I. To assess progression free survival (PFS) at 2 years after stem cell transplant (SCT) for high-risk hematologic malignancies receiving T-cell depleted grafts followed by escalating dose regimen (EDR) prophylactic DLI compared to historical controls not receiving DLI.

II. To assess the safety of EDR DLI for high-risk hematologic malignancies as measured by cumulative incidence of severe grade III-IV acute graft-versus-host disease (GVHD).

III. To measure outcomes of grade II-IV acute GVHD, non-relapse mortality, overall survival and chronic GVHD of EDR DLI.

IV. To assess the full donor chimerism rate in the CD3 compartment and immune reconstitution after EDR DLI.

OUTLINE:

Patients receive DLI intravenously (IV). Treatment repeats every 4-8 weeks for 5 doses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up periodically for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* INCLUSION CRITERIA PRIOR TO TRANSPLANT:
* The clinical trial will be offered to all high risk (defined 3 below) patients with hematologic malignancies who require stem cell transplants as part of their standard of care using matched related or unrelated donors
* Patients with high risk myeloid or lymphoid malignancies at stem cell transplant following American Society for Blood and Marrow Transplantation (ASBMT) criteria, including but not limited to conditions listed; these criteria apply BEFORE cyto-reductive therapy given within 28 days of planned conditioning:

  * Refractory acute myelogenous or lymphoid leukemia
  * Relapsed acute myelogenous or lymphoid leukemia
  * Myelodysplastic syndromes with 5% or more blasts
  * Chronic myelogenous leukemia in chronic phase 3 or more, blast phase presently, or second accelerated phase
  * Recurrent or refractory malignant lymphoma or Hodgkin's disease with less than a partial response at transplant
* High risk chronic lymphocytic leukemia defined as no response or stable disease to the most recent treatment regimen
* DONORS: Matched related or unrelated donor stem cell transplant (SCT) matched at human leukocyte antigen (HLA) A- B, C, and DRB1 by molecular methods; 7 of 8 matched donor acceptable for related donors
* T-cell depletion with anti-thymocyte globulin (ATG) (rabbit or horse) or at least 30 mg of alemtuzumab total in the conditioning regimen
* Immune suppression; planned post-transplant immune suppression should include tacrolimus or cyclosporin monotherapy (i.e., calcineurin inhibitor or CN) for alemtuzumab regimens and a second immune suppressant for ATG treated patients; other agents may be used if CN intolerance or toxicity occurs post-transplant
* Zubrod performance status (PS) 0-2 or equivalent Karnofsky PS
* Eligible for allogeneic transplant in the treating physicians' judgment and by institutional standards
* ELIGIBILITY TO RECEIVE DLI POST-TRANSPLANT:
* Donor lymphocytes available or able to be collected
* No evidence of disease by standard morphology; minimal residual disease or molecular evidence of disease will not exclude
* Absolute neutrophil count >= 500/μl
* Platelet count >= 20,000/μl without transfusion for 7 days
* Serum glutamic oxaloacetic transaminase (SGOT) and serum glutamate pyruvate transaminase (SGPT) =< 5 x upper limit of normal (ULN)
* Bilirubin =< 3 x ULN
* No evidence of grade II or higher acute GVHD or chronic GVHD at initiation of first DLI
* No systemic corticosteroids or immunosuppressive drugs (topical acceptable); replacement steroids for adrenal insufficiency are not excluded

Exclusion Criteria:

* EXCLUSION CRITERIA PRIOR TO TRANSPLANT:
* Pregnant or lactating females
* Hepatitis B with positive viral load prior to transplant conditioning or hepatitis C virus
* Human immune deficiency virus
* Psychiatric illness that may make compliance to the clinical protocol unmanageable or may compromise the ability of the patient to give informed consent
* Creatinine >= 2.0 mg/dL
* SGOT and SGPT >= 5 x ULN; liver biopsy preferred for such patients
* Bilirubin >= 3 x ULN (unless Gilbert's syndrome)
* Diffusing capacity of the lung for carbon monoxide (DLCO) < 50% corrected for hemoglobin
* Left ventricular ejection fraction or shortening fraction < 40%
* Unlikely to be able to procure additional donor lymphocytes

Ages: 14 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2013-04-04 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hongtao Liu, Principal Investigator — University of Chicago Comprehensive Cancer Center
Locations (1):
- University of Chicago Comprehensive Cancer Center, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (DLI)
Started | 77
Completed | 36
Not Completed | 41
Not completed — Death | 9
Not completed — Physician Decision | 17
Not completed — Relapse | 12
Not completed — GVHD | 2
Not completed — Graft Failure | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (DLI)
Number analyzed (Participants) | 77
Age, Continuous [Median (Full Range); unit: years] | 53 [20 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 51
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 70
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Who Are Able to Receive at Least One DLI Treatment
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (DLI)
Number analyzed (Participants) | 77
Participants | 36

2. Secondary Outcome: Progression Free Survival (PFS)
Description: Time to relapse or death as a result of any cause was evaluated at 2 years and the progression free survival rate was reported.
Time Frame: 2 years
Population: Patients received at least one DLI Treatment.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Treatment (DLI)
Number analyzed (Participants) | 36
percentage of patients | 43 [29 to 63.9]

3. Secondary Outcome: Overall Survival (OS)
Description: Computed using the Kaplan-Meier product-limit estimate and expressed as probabilities with a 95% CI.
Time Frame: At 2 years
Population: Patients received at least one DLI Treatment.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Treatment (DLI)
Number analyzed (Participants) | 36
percentage of patients | 59.7 [44.8 to 79.4]

4. Secondary Outcome: Rate of Acute GVHD (aGVHD) With Any Grade
Description: Estimated by cumulative incidence method.
Time Frame: At 1 year and 2 year
Population: Patients received at least one DLI Treatment.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Treatment (DLI)
Number analyzed (Participants) | 36
percentage of patients
  At 1 year | 41.8 [24.6 to 58.1]
  At 2 year | 41.8 [24.6 to 58.1]

5. Secondary Outcome: Rate of Chronic GVHD (cGVHD)
Description: Estimated by cumulative incidence method.
Time Frame: At 1 year and 2 year
Population: Patients received at least one DLI treatment.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Treatment (DLI)
Number analyzed (Participants) | 36
percentage of patients
  At 1 year | 26.6 [12.2 to 43.4]
  At 2 year | 26.6 [12.2 to 43.4]

6. Secondary Outcome: Treatment-related Mortality
Description: Estimated by cumulative incidence method. Cumulative incidence of treatment-related mortality with relapse of the original disease as the competing risk will be calculated.
Time Frame: At 2 year
Population: Patients received at least one DLI treatment.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Treatment (DLI)
Number analyzed (Participants) | 36
percentage of patients | 12.1 [3.7 to 25.9]

ADVERSE EVENTS:
Time Frame: 2 year
Arm/Group | Treatment (DLI)
All-Cause Mortality (participants affected / at risk) | 17/36
Serious Adverse Events (participants affected / at risk) | 12/36
Other Adverse Events (participants affected / at risk) | 1/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (DLI) (N=36)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Death (General disorders) | 2
Diarrhea from drug (Gastrointestinal disorders) | 1
Dizziness (Nervous system disorders) | 1
Fever (General disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 1
nervous system disorder (Nervous system disorders) | 1
Pneumonia (Reproductive system and breast disorders) | 1
Burn (Injury, poisoning and procedural complications) | 1
Acute Kindey Injury (Renal and urinary disorders) | 1
Small Bowel obstruction (Renal and urinary disorders) | 1
Hypotension (Vascular disorders) | 1
Disseminated zoster (Immune system disorders) | 1
Infection (Infections and infestations) | 1
leg fracture due to fall (Injury, poisoning and procedural complications) | 1
Liver GVHD (Investigations) | 2
Viral diarrhea (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (DLI) (N=36)
Sepsis (Infections and infestations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-12): https://cdn.clinicaltrials.gov/large-docs/16/NCT01839916/Prot_SAP_000.pdf